CLINICAL TRIAL: NCT01929616
Title: Regorafenib Assessment in Refractory Advanced Colorectal Cancer
Brief Title: Regorafenib Assessment in Refractory Advanced Colorectal Cancer(RegARd-C)
Acronym: RegARd-C
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jules Bordet Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-005655-16 EUDRACT
Record Dates: First submitted 2013-07-28; First posted 2013-08-28 (Estimated); Last update posted 2019-06-25 (Actual); Status verified 2017-03

CONDITIONS: Advanced Chemorefractory Colorectal Adenocarcinoma
Keywords: adenocarcinoma, colorectal,regorafenib
MeSH Terms: conditions — Adenocarcinoma | interventions — regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Regorafenib (Experimental): A treatment cycle is defined as a 4 weeks period. Regorafenib will be administered once a day orally at a dose of 160 mg (4 tablets of 40 mg), for 3 weeks.
  Interventions: Drug: regorafenib

INTERVENTIONS:
Drug: regorafenib — Patients will receive 160 mg regorafenib 1/day 3 weeks out of 4.
  Other Names: stivarga (registred name)

SUMMARY:
The general objectives are to evaluate activity and the safety of regorafenib in a population of patients bearing advanced, refractory colorectal cancers and to explore the different downstream molecular pathways to identify tumor response and resistance mechanisms.

DETAILED DESCRIPTION:
The primary objective is to identify in a population of patients bearing advanced, refractory colorectal cancers, those who draw no benefit from treatment with regorafenib. There is no specific hypothesis underlying sample size and the study is therefore to be seen as exploratory.

Secondary objectives:

* To analyze PFS and response rate (RR) in relationship with the same covariates as for OS
* To assess regorafenib efficacy (OS, PFS, RR) and safety profile in this study population.
* To assess the Disease control rate (DCR = Complete response [CR] + partial response [PR] + stable disease [SD])
* To compare the relative benefit (OS, PFS) of regorafenib according to history of treatment with bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven colorectal adenocarcinoma that is metastatic or unresectable and for which standard treatments do not exist or are no longer effective.
2. Age ≥ 18 years.
3. Life expectancy of greater than 12 weeks.
4. ECOG performance status ≤ 1.
5. Participants must have normal organ and bone marrow function as defined below:

   * Leukocytes >3,000/mcL,with an absolute neutrophil count >1,500/mcL, platelets >100,000/mcL, Hb >or=9g/dl.
   * Total bilirubin≤1.5×institutional ULN.
   * AST/ALT/P-Alk levels ≤ 2.5 × institutional ULN (≤5x institutional ULN in case of liver metastatic involvement).
   * Lipase ≤1.5 institutional ULN.
   * coagulation tests ≤ 1.5 x institutional ULN.
   * Creatinine ≤ 1.5× institutional ULN or creatinine clearance >30mL/min according to the Modified Diet in Renal Disease (MDRD) abbreviated formula.
6. Women of childbearing potential and men must agree to use adequate contraception prior to study entry, until at least 3 months after the last study drug administration.
7. Signed Written Informed Consent (IC).
8. Presence of a previously collected or freshly obtained at the time of study entry frozen metastatic tumor biopsy in a FDG-PET targetable lesion.
9. Presence of at least one metabolically measurable tumoral lesion on FDG PET-CT

Exclusion Criteria:

1. Prior treatment with sorafenib or regorafenib
2. Patients with previous cancer that is not disease-free for at least for 5 years prior to registration, EXCEPT for curatively treated cervical cancer in situ, non-melanoma skin cancer and superficial bladder tumors [Ta (Non-invasive tumor), Tis (Carcinoma in situ) and T1 (Tumor invades lamina propria)].
3. Participants who have had a major surgery, chemotherapy or radiotherapy within 4 weeks prior to entering the study.
4. Unresolved toxicity higher than NCI-CTCAE (version 4.0) Grade 1 attributed to any prior therapy/procedure excluding alopecia and oxaliplatin induced neurotoxicity ≤Grade 2.
5. Participants receiving any experimental agents.
6. Participants with known brain metastases.
7. Bleeding diathesis, history of cardiovascular ischemic disease or cerebrovascular incident within the last six months.
8. Any hemorrhage or bleeding event NCI-CTCAE v.4 Grade >or= 3 within 4 weeks prior to the start of study medication.
9. Uncontrolled concurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure (New York Heart Association (NYHA)class> or=2), unstable angina pectoris, cardiac arrhythmia requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted).
10. Uncontrolled hypertension.
11. Patients with seizure disorder requiring medication.
12. Any history of organ allograft.
13. Pleural effusion or ascites affecting respiration.
14. Uncontrolled diabetes.
15. Non-healing wound, ulcer, or bone fracture.
16. Known history of human immunodeficiency virus (HIV) infection, or active hepatitis B or C, or chronic hepatitis B or C requiring treatment with antiviral therapy.
17. Interstitial lung disease with ongoing signs and symptoms.
18. Renal failure requiring hemo-or peritoneal dialysis.
19. Dehydration NCI-CTCAE v.4 grade >1.
20. Medical,psychological or social conditions that may interfere with the patient's ability to understand informed consent and participation in the study or evaluation of the study results.
21. Known hypersensitivity to the study drug or excipients in the formulation.
22. Any illness or medical conditions that are unstable or could jeopardize the safety of the patient and his/her compliance in the study.
23. Pregnant or lactating women.
24. Subjects unable to swallow oral medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2013-08; Primary Completion 2016-05-13 (Actual); Study Completion 2019-06-17 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | 2 years from first patient in

SECONDARY OUTCOMES:
Occurence of Adverse events | Every 28 days till 28 days after stopping therapy. An average of 2 months is expected.
  Assessment of safety will follow the WHO guidelines and classified according to NCI-CTCAE v. 4.0 and will be performed every 28 days until 28 days (safety follow up visit) after stopping therapy. Reasons for stopping therapy may include progression of disease or unbearable toxicities, or patient's decision.
Evaluation of tumour response | Every 2 months till progression of the disease. An average of 2 months is expected.
  RECIST 1.1-based radiological assessment (CT or MRI) will be made every 2 cycles, starting at day 28 of the second cycle till demonstration of progressive disease. An average of 2 months is expected.
Metabolic response assessed by FDG PET | 2 FDGPET will be perfomed : at Baseline (day 0) and at D14
  FDGPET will be done twice during the study course : at baseline (at day 0, before treatment begin) and after 2 weeks.
Molecular aberrations | at day 0 (before treatment begins) and at D14, then repeated every 2 months until progression. An average of 2 months is expected.
  Genetic, epigenetic and molecular aberrations will be investigated using gene expression profiling, RNA and exome sequencing, and methylation profiling on the tumor biopsies and repeated blood samples collected during the trial. The relationship between the molecular aberrations,the patient's outcome (PFS, OS) and with metabolic response after treatment with regorafenib will be studied.

CONTACTS AND LOCATIONS:
Overall Officials: Alain Hendlisz, MD, Study Chair — Jules Bordet Institute
Locations (17):
- Belgium (17):
  - UZA, Antwerp, Edegem
  - Jules Bordet Institute, Brussels
  - Hopital Erasme, Brussels
  - Cliniques Universitaires Saint Luc, Brussels
  - Grand Hopital de Charleroi, Charleroi
  - UZ Ghent, Ghent
  - AZ groeninge, Kortrijk
  - Centre Hospitalier Universitaire de Liège, Liège
  - Clinique St Joseph, Liège
  - Centre hospitalier de Jolimont, Lobbes
  - CHU Ambroise Paré, Mons
  - Centre Hospitalier Régional de Namur, Namur
  - Clinique et Maternité Sainte Elisabeth, Namur
  - Clinique Saint Pierre, Ottignies
  - Hartziekenhuis Roeselare-Menen (HHRM), Roeselare
  - AZ Turnhout, Turnhout
  - Cliniques Universitaires UCL de Mont-Godinne, Yvoir

REFERENCES:
- [Derived] Charette N, Vandeputte C, Ameye L, Bogaert CV, Krygier J, Guiot T, Deleporte A, Delaunoit T, Geboes K, Van Laethem JL, Peeters M, Demolin G, Holbrechts S, Flamen P, Paesmans M, Hendlisz A. Prognostic value of adipose tissue and muscle mass in advanced colorectal cancer: a post hoc analysis of two non-randomized phase II trials. BMC Cancer. 2019 Feb 12;19(1):134. doi: 10.1186/s12885-019-5319-8. PMID 30744591
- [Derived] Hendlisz A, Deleporte A, Vandeputte C, Charette N, Paesmans M, Guiot T, Garcia C, Flamen P. Regorafenib assessment in refractory advanced colorectal cancer: RegARd-C study protocol. BMJ Open. 2015 Mar 9;5(3):e007189. doi: 10.1136/bmjopen-2014-007189. PMID 25753361